CLINICAL TRIAL: NCT03767543
Title: A Randomized, 26-week, Open-label, 2-treatment Arm, Parallel Group Multicenter Study Comparing the Efficacy and Safety of Insulin Glargine/Lixisenatide Fixed-ratio Combination (Soliqua™) Titrated Using a Simple Titration Algorithm (One Unit Daily Adjustment) Compared With Insulin Glargine/Lixisenatide Fixed-ratio Combination (Soliqua™) Titrated by Weekly Adjustment in Patients With Type 2 Diabetes Mellitus (T2DM)
Brief Title: Study Comparing the Efficacy and Safety of Insulin Glargine (Basal Insulin)/Lixisenatide (GLP-1 Receptor Agonist) Combination (Soliqua™) in Patients With Type 2 Diabetes Mellitus (T2DM)
Acronym: LixilanOne CAN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LPS15544; U1111-1215-0238 (Other: UTN)
Record Dates: First submitted 2018-12-05; First posted 2018-12-06 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- iGlarlixi DAILY (Experimental): Titration Group 1: Addition of 1 unit per day until pre-stated fasting self-monitoring plasma glucose (SMBG) level is reached
  Interventions: Drug: INSULIN GLARGINE/LIXISENATIDE HOE901/AVE0010
- iGlarlixi WEEKLY (Active Comparator): Titration Group 2: Algorithm of weekly adjustment until pre-stated fasting self-monitoring plasma glucose (SMBG) level is reached
  Interventions: Drug: INSULIN GLARGINE/LIXISENATIDE HOE901/AVE0010

INTERVENTIONS:
Drug: INSULIN GLARGINE/LIXISENATIDE HOE901/AVE0010 — Pharmaceutical form: Solution for injection Route of administration: Subcutaneous

SUMMARY:
Primary Objective:

To demonstrate that the simple daily titration algorithm is non-inferior to the weekly titration algorithm according to Canadian labeling.

Secondary Objective:

To gain additional information on the efficacy and safety of using a simple patient-titration protocol for administration of insulin glargine/lixisenatide fixed-ratio combination (iGlarLixi).

DETAILED DESCRIPTION:
The maximum duration of study per patient is approximately 29 weeks including a 2-week screening, a 26-week randomized active-controlled treatment period, and 3-day post-treatment safety follow-up period.

ELIGIBILITY:
Inclusion criteria:

* Adult subject ≥ 18 years
* Patients with type 2 diabetes mellitus (T2DM) based on Diabetes Canada 2018 Clinical Practice Guidelines criteria and diagnosed at least 6 months prior to the screening visit
* Uncontrolled glycemia with an A1c ≥7.5% and ≤10.5%
* Patients treated for at least 6 months on any basal insulin (including but not limited to insulin glargine, Toujeo®, Degludec®, etc.) ± oral anti-diabetic drug (OADs)
* The total basal insulin dose must be ≤ 40 units/day
* The OADs allowed at inclusion are metformin, insulin secretagogues, dipeptidyl-peptidase-4 inhibitors (DPP4) inhibitors and SGLT2 inhibitors; with no change in OAD dose for at least 2 months prior to randomization
* Body mass index (BMI) between 20 kg/m2 and 40 kg/m2 inclusively

Exclusion criteria:

* History of severe hypoglycemia or hypoglycemia unawareness
* History of metabolic acidosis, including diabetic ketoacidosis within 1 year prior to screening visit
* Current or previous (known intolerance to GLP-1s) treatment with glucagon like peptide-1 (GLP-1) receptor agonist
* Current use of rapid-acting insulin or premix insulins or use of these insulins within 3 months prior to the screening visit
* Use of systemic glucocorticoids (excluding topical and inhaled forms) for a total duration of 1 week or more within 3 months prior to the screening visit
* Use of weight loss drugs within 3 months prior to the screening visit
* Patients with conditions/concomitant diseases that will affect safe participation in this study (e.g. active malignant tumor, major systemic diseases, presence of clinically significant diabetic retinopathy or presence of macular edema likely to require treatment within the study period, etc.)
* Women of childbearing potential (WOCBP) not protected by an effective contraceptive method of birth control and/or who are unwilling or unable to be tested for pregnancy
* Positive serum pregnancy test in WOCBP, pregnancy or lactation
* Clinically relevant history of gastrointestinal disease associated with prolonged nausea and vomiting, including (but not limited to): gastroparesis, unstable (i.e. worsening) or uncontrolled (i.e. prolonged nausea and vomiting) gastroesophageal reflux disease requiring medical treatment within 6 months prior to the time of screening visit
* History of pancreatitis (unless pancreatitis was related to gallstones and treated with cholecystectomy), pancreatitis during previous treatment with incretin therapies, chronic pancreatitis, pancreatectomy, or stomach/gastric surgery
* Personal or immediate family history of medullary thyroid cancer or genetic conditions that predispose the patient to medullary thyroid cancer (e.g. multiple endocrine neoplasia syndromes)

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 265 (Actual)
Dates: Start 2019-03-11 (Actual); Primary Completion 2020-10-23 (Actual); Study Completion 2020-10-23 (Actual)

PRIMARY OUTCOMES:
Change in glycated hemoglobin (HbA1c)% | Baseline to Week 26
  Absolute mean change in HbA1c from baseline to Week 26; HbA1c is expressed in % (unit)

SECONDARY OUTCOMES:
Percentage of patients achieving HbA1c ≤7% at Week 26 | At Week 26
  Percentage of patients achieving A1c ≤7%
Change in fasting plasma glucose (FPG) from baseline to Week 12 | Baseline to Week 12
  Change in FPG from baseline to Week 12
Change in FPG from baseline to Week 26 | Baseline to Week 26
  Change in FPG from baseline to Week 26
Change in fasting self-monitoring plasma glucose (SMPG) from baseline to Week 12 | Baseline to Week 12
  Change in fasting SMPG from baseline to Week 12
Change in fasting SMPG from baseline to Week 26 | Baseline to Week 26
  Change in fasting SMPG from baseline to Week 26
Change in 7-point SMPG profile from baseline to Week 12 | Baseline to Week 12
  Change in 7-point SMPG profile from baseline to Week 12
Change in 7-point SMPG profile from baseline to Week 26 | Baseline to Week 26
  Change in 7-point SMPG profile from baseline to Week 26
Change in body weight from baseline to Week 26 | Baseline to Week 26
  Change in body weight (kg)
Percentage of patients achieving A1c ≤7% with no body weight gain and/or hypoglycemia (severe or documented symptomatic (≤3.9 mmol/L) at Week 26 | Baseline to Week 26
  Composite endpoint expressed as percentage of patients A1c ≤7% with no body weight gain and/or hypoglycemia (severe or documented symptomatic (≤3.9 mmol/L)
Insulin glargine dose | At Week 26
  Insulin glargine dose (expressed in units)
Percentage of patients requiring rescue therapy | Baseline to Week 26
  Percentage of patients requiring rescue therapy during the 26-week open-label treatment period
Percentage of patients experiencing at least 1 hypoglycemia episode (≤3.9 mmol/L) over 26 weeks | Baseline to Week 26
  Percentage of patients experiencing at least 1 hypoglycemia episode defined as ≤3.9 mmol/L
Percentage of patients experiencing at least 1 hypoglycemia episode (<3.0 mmol/L) over 26 weeks | Baseline to Week 26
  Percentage of patients experiencing at least 1 hypoglycemia episode defined as <3.0 mmol/L
Annualized rate of hypoglycemia (≤3.9 mmol/L) over 26 weeks | Baseline to Week 26
  Mean number of hypoglycemia episodes (≤3.9 mmol/L) per patient year of exposure over 1 year
Annualized rate of hypoglycemia (<3.0 mmol/L) over 26 weeks | Baseline to Week 26
  Mean number of hypoglycemia episodes (<3.0 mmol/L) per patient year of exposure over 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (32):
- Canada (32):
  - Investigational Site Number 1240004, Barrie
  - Investigational Site Number 1240006, Brampton
  - Investigational Site Number 1240002, Brampton
  - Investigational Site Number 1240005, Burlington
  - Investigational Site Number 1240003, Calgary
  - Investigational Site Number 1240024, Chicoutimi
  - Investigational Site Number 1240014, Concord
  - Investigational Site Number 1240017, Etobicoke
  - Investigational Site Number 1240030, Greenfield Park
  - Investigational Site Number 1240031, Halifax
  - Investigational Site Number 1240026, Hamilton
  - Investigational Site Number 1240011, Laval
  - Investigational Site Number 1240016, London
  - Investigational Site Number 1240015, London
  - Investigational Site Number 1240019, Mirabel
  - Investigational Site Number 1240018, Montreal
  - Investigational Site Number 1240023, Montreal
  - Investigational Site Number 1240020, Montreal
  - Investigational Site Number 1240029, Montreal
  - Investigational Site Number 1240027, Nepan
  - Investigational Site Number 1240025, Newmarket
  - Investigational Site Number 1240021, Oakville
  - Investigational Site Number 1240009, Oshawa
  - Investigational Site Number 1240008, Québec
  - Investigational Site Number 1240022, Québec
  - Investigational Site Number 1240028, Saint-Lambert
  - Investigational Site Number 1240013, Saint-Marc-des-Carrieres
  - Investigational Site Number 1240033, Toronto
  - Investigational Site Number 1240001, Toronto
  - Investigational Site Number 1240012, Vancouver
  - Investigational Site Number 1240007, Victoriaville
  - Investigational Site Number 1240032, Winnipeg

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Yale JF, Roborel de Climens A, Aggarwal N, Dex T, Gerstein HC, Harris S, Hramiak I, Stewart J, Leiter LA. Ease of Use of the iGlarLixi SoloStar Pen from the LixiLan ONE CAN Pen Sub-Study: Questionnaire Findings from People Living with Type 2 Diabetes and Their HealthCare Providers. Diabetes Ther. 2023 Feb;14(2):377-386. doi: 10.1007/s13300-022-01353-6. Epub 2022 Dec 27. PMID 36574199
- [Derived] Hramiak I, Gerstein HC, Leiter LA, Yale JF, Bajaj HS, Stewart J, Toutounji MJ, Harris SB. Comparing a daily versus weekly titration algorithm in people with type 2 diabetes switching from basal insulin to iGlarLixi in the LixiLan ONE CAN randomized trial. Diabetes Obes Metab. 2022 Oct;24(10):1998-2007. doi: 10.1111/dom.14787. Epub 2022 Jun 29. PMID 35670659